CLINICAL TRIAL: NCT05701319
Title: Left Main Intervention in Myocardial Infarction and Acute Coronary Syndromes The LIMACS Multicenter Registry
Brief Title: Left Main Intervention in Myocardial Infarction and Acute Coronary Syndromes
Acronym: LIMACS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Collaborators: Tanta University (Other); Al-Azhar University (Other); Egyptian Soceity of Cardiology (Unknown)
Responsible Party: Principal Investigator, Salma Taha, Ass.Professor of Cardiology, Assiut University
Other Study IDs: LM in ACS
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: LMN Disease
Keywords: UPLM; ACS; PPCI
MeSH Terms: conditions — Motor Neuron Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: PCI — percutaneous coronary intervention

SUMMARY:
Limited data have been published on the management and outcome of patients with acute coronary syndrome (ACS) undergoing percutaneous coronary intervention (PCI) that involves the left main (LM) coronary artery. Little is known about different strategies and techniques of percutaneous revascularization and long-term outcomes of these patients. Beside scarcity of data, most studies represent outmoded experience not reflecting contemporary advances in stent technologies, with the introduction of newer generation thinner strut drug eluting stents (DES), bioresorbable polymers, and faster re-endothelization properties promoting vascular healing and endothelial repair. These advances have significantly reduced the rate of ischemic (especially thrombotic) complications in different cohorts. Whether these advances would alter the outcome of PCI that involves the LM in patients with ACS is yet to be explored.

II. Objective

1. To explore real-world PCI strategies and techniques in patients with unprotected LM coronary disease presenting with ACS
2. To explore short- and long-term outcomes of patients of ACS with LM intervention III. Study endpoints Primary endpoint Major adverse cardiovascular events (MACE) at one year; a composite of all-cause mortality, non-fatal myocardial infarction (MI), or unplanned revascularization* *With further extended yearly follow-up to 5 years Secondary endpoints

1) All-cause death at one year* 2) Non-fatal MI at one year* 3) Any unplanned revascularization at one year* 4) Target vessel revascularization (TVR) at one year* 5) Academic Research Consortium (ARC) definite/probable stent thrombosis at one year* 6) Bleeding Academic Research Consortium (BARC) type 3 or 5 bleeding at one year* 7) Contrast induced nephropathy (CIN) defined as serum creatinine rise >25% or absolute increase >0.5 mg/dL within 72 hours after index PCI 8) Echocardiographic left ventricular ejection fraction (LVEF)% [Time Frame: from 6 to 12 months after index PCI]* 9) Angiographic (re)stenosis of the LM [Time Frame: from 6 to 12 months after index PCI] (Optional)

DETAILED DESCRIPTION:
IV. Study Type Single-arm, prospective and retrospective, multicenter, open-label registry V. Study Population Consecutive adult patients admitted with ACS (diagnosed within 72 hours before hospitalization) undergoing revascularization will be screened and considered for inclusion in the study. Patients with ACS (MI or unstable angina) undergoing PCI that involves unprotected LM with a DES will be enrolled; either same-session (during index procedure, with culprit lesion PCI) or scheduled in-hospital (same hospitalization with index PCI).

Exclusion criteria:

* Cannot provide informed consent
* Un-able/willing to comply with the study requirements including follow up visits
* Life expectancy <1 year
* Contraindications to anti-platelet drugs
* Rescue PCI (PCI after failed thrombolytic therapy)
* Prior CABG (patent LIMA)
* Severe CKD (GFR<30 ml/min) VI. Study Treatment Eligible patients will receive ASA as per standard of care and ticagrelor/clopidogrel loading dose according to recent guidelines.

In patients with multivessel disease, treatment only of the culprit lesion/target vessel during index PCI is recommended. Clinical follow up (clinic visit/phone call) will be scheduled at 1, 6, 12, and 60 months. Control invasive coronary angiography at 6-12 months after index PCI will be encouraged. Echocardiographic evaluation of LVEF is recommended at 6 and 12 month-follow up.

VII. Study Duration Enrollment Duration: 24 months Follow up duration: Five years (predefined follow up scheduled at 1, 6, 12, and 60 months). Annual follow up between 12 and 60 months are encouraged but not mandated.

VIII. Estimated Enrollment 500 patients

Sample Size Calculation: As this is a single-arm registry, sample size calculation is not mandatory. However, a sample size of 450 subjects would be required according to the following assumptions:

Expected event rate: 3.0%, test significance level (alpha): 2.5% (1-sided), sample size: 400, power: 80%, expected drop out/protocol violation: 10%, final sample size: 450.

IX. Prespecified Subgroup Analyses

1. One vs. two-stent LM-bifurcation technique
2. LM culprit vs. non-culprit intervention
3. Multivessel vs. single-vessel disease
4. Complete vs. incomplete revascularization
5. Diabetes mellitus (yes/no)
6. STEMI: primary vs. scheduled pharmaco-invasive PCI X. Projected Study Timelines

   * First patient enrollment: January 2023
   * Last patient enrollment: December 2024
   * First 12-month FUP: January 2024
   * Last 12-month FUP: December 2025 (1ry endpoint completion)
   * Final 5-year FUP: December 2028 (Study conclusion)

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients admitted with ACS (diagnosed within 72 hours before hospitalization) undergoing revascularization will be screened and considered for inclusion in the study.

Patients with ACS (MI or unstable angina) undergoing PCI that involves unprotected LM with a DES will be enrolled; either same-session (during index procedure, with culprit lesion PCI) or scheduled in-hospital (same hospitalization with index PCI).

Exclusion Criteria:

* cannot provide informed consent
* Un-able/willing to comply with the study requirements including follow up visits
* Life expectancy <1 year
* Contraindications to anti-platelet drugs
* Rescue PCI (PCI after failed thrombolytic therapy)
* Prior CABG (patent LIMA)
* Severe CKD (GFR<30 ml/min)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients with ACS and LM disease
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | one year
  a composite of all-cause mortality, non-fatal myocardial infarction (MI), or unplanned revascularization*

SECONDARY OUTCOMES:
All-cause death | one year
  death due to any cause
Non-fatal MI | one year
  Myocardial infarction
Any unplanned revascularization | one year
  revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Osama Shoaib, lecturer, Principal Investigator — Tanta University
Locations (3):
- Egypt (3):
  - Assiut University, Asyut
  - Alazhar university, Cairo
  - Tanta University, Tanta

IPD SHARING:
Plan to Share IPD: Undecided
through google drive